CLINICAL TRIAL: NCT02537756
Title: Developing a Self-persuasion Intervention Promoting Adolescent HPV Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Southern Methodist University (Other); Parkland Health and Hospital System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: STU 022013-016; 1R01CA178414-01 (NIH)
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Human Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1- Verbalize, Choice (Experimental): Parents will use a tablet-based application (Project Voice) that directs them to verbalize their own arguments based on topics they choose
  Interventions: Behavioral: Project Voice
- 2- Listen, Choice (Experimental): Parents will use a tablet-based application (Project Voice) that directs them to listen to peer-generated arguments based on topics they choose
  Interventions: Behavioral: Project Voice
- 3- Verbalize, Assigned (Experimental): Parents will use a tablet-based application (Project Voice) that directs them to verbalize their own arguments based on topics assigned to them
  Interventions: Behavioral: Project Voice
- 4- Listen, Assigned (Experimental): Parents will use a tablet-based application (Project Voice) that directs them to listen to peer-generated arguments based on topics assigned to them
  Interventions: Behavioral: Project Voice

INTERVENTIONS:
Behavioral: Project Voice — A tablet-based intervention that directs participants through different activities related to adolescent HPV vaccination based on their assigned condition

SUMMARY:
HPV vaccine coverage among adolescents in the US is suboptimal. This is particularly true among traditionally underserved adolescents. Few parent-targeted interventions have focused on the parental decision-making process. Self-persuasion, generating one's own arguments for engaging in a behavior, may be an effective means to influence parents' motivation to vaccinate their children. In a three-phase study, investigators are using quantitative and qualitative research methods to develop and refine a tablet-based self-persuasion intervention for parents who are undecided about the HPV vaccine. This clinical trial submission focuses on the second phase of the study. The results of the second phase will inform the third phase of the trial (also registered in clinical trials).

DETAILED DESCRIPTION:
Despite the fact that HPV vaccination is recommended for male and female adolescents, HPV vaccine 3 dose coverage among adolescents is poor (38% for girls, 14% for boys). HPV-related cancers are a significant burden on the US healthcare system and could be prevented through adolescent vaccination. Rates of vaccination are suboptimal among underserved populations (uninsured, low-income, racial and ethnic minorities) often seen in safety-net clinics. Few interventions have been designed that target decision-making among parents of unvaccinated adolescents. Self-persuasion, generating of one's own arguments for a health behavior, may be an effective means of influencing HPV vaccination behaviors among undecided or ambivalent parents. Through three stages, investigators will identify and develop a self-persuasion intervention strategy to promote adolescent HPV vaccination in safety-net clinics. The current trial, Stage 2, is a four-arm randomized controlled trial (RCT), using a 2x2 factorial design, in which investigators will assign participants to one of four self-persuasion intervention conditions that vary by cognitive processing level (verbalize vs. listen to arguments) and choice of argument topics (parents choose vs. are assigned topics) to identify which intervention condition is optimal. Conducted in a laboratory setting, investigators will identify and select the optimal intervention condition through quantitative analysis of the effects on parents' vaccination intentions and qualitatively by exploring parental experiences with the self-persuasion tasks.

ELIGIBILITY:
Inclusion Criteria:

* Undecided parents (18 years and older) whose children are 11-17 year old patients who have not begun the HPV vaccine series.

Exclusion Criteria:

* Parents whose child is a pregnant adolescent
* Lack telephone access
* Having impairing hearing or speech
* Participants will be excluded from participation in future stages

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2019-10-26 (Actual)

PRIMARY OUTCOMES:
Survey Items Measuring Parental Intentions to vaccinate | During the intervention visit (1 hr)
  Change in intentions of the parent to vaccinate from baseline survey to exit survey using measures adapted from Gerend & Shepherd (2012). Intentions Likert Scale responses range from 1-very likely to 5-very unlikely.

SECONDARY OUTCOMES:
HPV vaccination behavior documented in the electronic medical record, initiation | 12 months
  Number of parents who initiated the series by vaccinating their child within 12 months of the study appointment as evidenced by documentation in the child's electronic medical record.
Change in Decision Stage | During the intervention visit (1 hr)
  Change in decision stage response of parents from baseline survey to post-educational video to post-intervention tasks.

OTHER OUTCOMES:
HPV vaccination behavior documented in the electronic medical record, completion | 15 months
  Number of doses received and the dates of those doses within 15 months of the study appointment as evidenced by documentation in the child's electronic medical record.
Vaccination Concerns, qualitative | During the intervention visit (1 hr)
  Number of parents reporting concerns during the intervention and exit interview; Describe the theme/category of concern expressed by parents about HPV vaccination
Manipulation checks | During the intervention visit (1 hr)
  Measure of the accuracy of parental argument recall during intervention (cognitive processing: verbalize own arguments); Change in autonomous motivation during intervention (argument topic choice).

CONTACTS AND LOCATIONS:
Overall Officials: Jasmin A Tiro, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Austin S Baldwin, PhD, Principal Investigator — Southern Methodist University
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (including data dictionaries) will be made available, in addition to study protocols, the statistical analysis plan, and the informed consent form. The data will be made available upon publication to researchers who provide a methodologically sound proposal and sign a data use agreement. Proposals should be submitted to Dr. Jasmin Tiro (jasmin.tiro@utsouthwestern.edu).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2020, for 10 years
Access Criteria: Researchers who provide a methodologically sound proposal and sign a data use agreement. Proposals should be submitted to Dr. Jasmin Tiro (jasmin.tiro@utsouthwestern.edu).

REFERENCES:
- [Derived] Tiro JA, Lee SC, Marks EG, Persaud D, Skinner CS, Street RL, Wiebe DJ, Farrell D, Bishop WP, Fuller S, Baldwin AS. Developing a Tablet-Based Self-Persuasion Intervention Promoting Adolescent HPV Vaccination: Protocol for a Three-Stage Mixed-Methods Study. JMIR Res Protoc. 2016 Jan 29;5(1):e19. doi: 10.2196/resprot.5092. PMID 26825137